CLINICAL TRIAL: NCT05693103
Title: The Effect of High-Intensity Focused Electromagnetic on Urinary Incontinence Symptoms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-F(I)-20210133
Record Dates: First submitted 2022-12-21; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: Urinary Incontinence, Stress Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Urinary Incontinence: Stress Urinary Incontinence Urge incontinence
  Interventions: Device: High-Intensity Focused Electromagnetic therapy

INTERVENTIONS:
Device: High-Intensity Focused Electromagnetic therapy — The HPM-6000UF is a non-invasive therapeutic device. The device produces electromagnetic field that interacts with the tissues of the human body.
  The electromagnetic field delivered in the muscular or neuronal tissue area is triggering the stimulation and tonisation.
  Other Names: EMSELLA

SUMMARY:
This study is aimed at women's pelvic floor muscles, especially urinary incontinence caused by pelvic floor muscle relaxation or pelvic prolapse, to observe whether the use of (HIFEM) high-intensity focused magnetic energy chairs can help the pelvic floor muscles after this treatment Strengthening to improve the symptoms of urinary incontinence caused by the compression of the sacral nerve plexus caused by the downward movement of the uterus, thereby improving the social life and quality of life of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Women over 20 years old.
2. Symptoms of urinary incontinence (including: stress incontinence, urge incontinence).
3. Blood tests confirmed that the number of platelets was 150,000-450,000/UL, and the coagulation function (PT) index was normal.

Exclusion Criteria:

1. Pregnant and lactating women.
2. Patients with acute or chronic cardiovascular disease.
3. Patients with acute or chronic infectious diseases.
4. Patients with malignant tumors, uterine fibroids, and gynecological cysts, who have been evaluated by doctors as unsuitable.
5. Those who have undergone lower abdominal or genital-related surgery and have been evaluated by doctors as unsuitable.
6. Patients with pulmonary insufficiency.
7. People with metal and electronic implants (such as: pacemaker, defibrillator, neurostimulator).
8. Those with bleeding disorders or receiving anticoagulant therapy.
9. Use drug pumps.
10. People with skin allergies or skin diseases.
11. Those unable to sign the subject's consent form.

Min Age: 20 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with stress urinary incontinence, urge incontinence.
Study Population: Collect 30 women with urinary incontinence symptoms (including: stress urinary incontinence, urge urinary incontinence)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Urodynamic study | One hour
  Urodynamic testing is any procedure that looks at how well parts of the lower urinary tract-the bladder, sphincters, and urethra-work to store and release urine. Most urodynamic tests focus on how well your bladder can hold and empty urine. Urodynamic tests can also show whether your bladder is contracting when it's not supposed to, causing urine to leak.
Questionnaire | fifteen minutes
  Female Sexual Function Index, International Consultation on Incontinence Questionnaire, Urogenital Distress Inventory-6, Incontinence Impact Questionnaire-7, The International Consultation on Incontinence, Pelvic Organ Prolapse Distress Inventory-6, Overactive Bladder Symptom Score, The global response assessment.
Physiological parameter | five minutes
  Age, BMI in kg/m^2, Pregnancy and childbirth, Year of Symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan